CLINICAL TRIAL: NCT05609162
Title: Effects of Local and Systemic Treatments in Brain Metastases With Poor Prognostic Factors: Multicenter Retrospective Study
Brief Title: Treatments for Brain Metastases With Poor Prognostic Factors
Acronym: TBMPPF
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Sun Yat-sen University (Other)
Collaborators: Cancer Hospital of Guangxi Medical University (Other); People's Hospital of Guangxi Zhuang Autonomous Region (Other); First Affiliated Hospital of Guangxi Medical University (Other)
Responsible Party: Principal Investigator, Yonggao Mou, Department of Neurosurgery, Sun Yat-sen University
Other Study IDs: B2020-218-01
Record Dates: First submitted 2022-11-02; First posted 2022-11-08 (Actual); Last update posted 2022-12-15 (Actual); Status verified 2022-12

CONDITIONS: Brain Metastases
Keywords: Brain Metastases; local treatments; systemic treatments; poor prognosis
MeSH Terms: conditions — Brain Neoplasms | interventions — Radiation; Drug Therapy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- local treatment group vs non-local treatment group: Participants underwent local treatments such as surgical resection or radiotherapy or surgical resection plus radiotherapy were divided into local treatment group or otherwise into non-local treatment group
  Interventions: Procedure: neurosurgical resection
- systemic treatment group vs non-systemic treatment group: Participants underwent systemic treatments such as chemotherapy or target therapy or chemotherapy plus target therapy were divided into systemic treatment group or otherwise into non-systemic treatment group
- local treatment group vs systemic treatment group: Participants underwent local treatments such as surgical resection or radiotherapy or surgical resection plus radiotherapy were divided into local treatment group; Participants underwent systemic treatments such as chemotherapy or target therapy or chemotherapy plus target therapy were divided into systemic treatment group
  Interventions: Procedure: neurosurgical resection
- local treatment group vs local treatment+systemic treatment group: Participants underwent local treatments such as surgical resection or radiotherapy or surgical resection plus radiotherapy were divided into local treatment group; Participants underwent local treatment plus systemic treatment were divided into local treatment+systemic treatment group
  Interventions: Procedure: neurosurgical resection
- systemic treatment group vs local treatment+systemic treatment group: Participants underwent systemic treatments such as chemotherapy or target therapy or chemotherapy plus target therapy were divided into systemic treatment group; Participants underwent local treatment plus systemic treatment were divided into local treatment+systemic treatment group
  Interventions: Procedure: neurosurgical resection
- local treatment+systemic treatment group vs non-local treatment+systemic treatment group: Participants underwent local treatment plus systemic treatment were divided into local treatment+systemic treatment group or otherwise into non-local treatment+systemic treatment group
  Interventions: Procedure: neurosurgical resection

INTERVENTIONS:
Procedure: neurosurgical resection — neurosurgical resection, stereotactic radiosurgery (SRS), whole brain radiotherapy(WBRT), EGFR target drugs, Immune checkpoint inhibitors，cisplatin, temozolomide
  Other Names: radiation; chemotherapy; target therapy
  Groups: local treatment group vs local treatment+systemic treatment group; local treatment group vs non-local treatment group; local treatment group vs systemic treatment group; local treatment+systemic treatment group vs non-local treatment+systemic treatment group; systemic treatment group vs local treatment+systemic treatment group

SUMMARY:
The goal of this observational study is to learn about treatments in brain metastases with poor prognostic factors. The main questions it aims to answer are:

* What kind of local treatment provides a survival benefit for patients with poor prognostic factors?
* What kind of systemic treatment provides a survival benefit for patients with poor prognostic factors?
* Will the combination of local treatment and systemic treatment provide a survival benefit for patients with poor prognostic factors?

Participants will be asked to provide personal information about their living status, symptoms, and disease control during the follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Evidence of pathological diagnosis of primary tumor;
2. Brain metastases confirmed by enhanced magnetic resonance imaging;
3. Complete clinical information

Exclusion Criteria:

1. Survival time less than 30 days;
2. If surgical treatment is accepted, the surgical treatment is not tumor resection, but ventricle puncture, biopsy and other non-tumor reducing surgery;
3. Incomplete clinical data;
4. Patients with 2 or more types of tumors.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Hospital clients from Sun Yat-sen University Cancer Center, Guangxi Medical University Cancer Hospital, The People's Hospital Of Guangxi Zhuang Autonomous Region, and the First Affiliated Hospital of Guangxi Medical University will be selected.
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2022-12-15 (Estimated); Primary Completion 2023-11-20 (Estimated); Study Completion 2024-11-20 (Estimated)

PRIMARY OUTCOMES:
OS | From date of first follow-up until the date of documented death from any cause, assessed up to 120 months
  Overall survival time

SECONDARY OUTCOMES:
PFS | From date of first follow-up until the date of first documented progression, assessed up to 120 months
  Progression-free survival time

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
We decided not to share the IPD because the study involved a lot of people's privacy

REFERENCES:
- [Derived] Li A, Feng D, Liu C, Huang C, Li T, Wei D, Wei F, Shen M, Qin C, Deng S, Liang H, Mo P, Dong M, Yu Y, Liang L. Prognostic Analysis of Lung Cancer With Brain Metastases in Elderly Patients: A Multicenter Retrospective Study. Aging Med (Milton). 2025 Dec 31;8(6):585-591. doi: 10.1002/agm2.70060. eCollection 2025 Dec. PMID 41531790